CLINICAL TRIAL: NCT03191240
Title: AMCPR (Augmented-Medication CardioPulmonary Resuscitation) for Improving Outcome in Patient With Cardiac Arrest: Multi-center, Double-blind, Prospective Randomized Clinical Trial.
Brief Title: AMCPR (Augmented-Medication CardioPulmonary Resuscitation) Trial for OHCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Won Young Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMCPR
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest; Vasopressin
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Diabetes Insipidus | interventions — Vasopressins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressins (Experimental): Additional vasopressin 40 IU intravenous injection for 2 times
  Interventions: Drug: Vasopressins
- Normal saline (Placebo Comparator): Additional normal saline intravenous injection for 2 times
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Vasopressins — Administer additional vasopressin 40 IU IV for 2 times during cardiopulmonary resuscitation
  Other Names: Vasopressin inj
  Arms: Vasopressins
Drug: Normal saline — Placebo
  Other Names: 0.9% sodium chloride
  Arms: Normal saline

SUMMARY:
The investigators aimed to evaluate the effect of AMCPR (Augmented-Medication CardioPulmonary Resuscitation: administration of additional vasopressin to titrate to arterial diastolic blood pressure over 20 mmHg) on cardiopulmonary resuscitation results and outcomes in out-of-hospital cardiac arrest patients.

DETAILED DESCRIPTION:
Non-traumatic out-of-hospital cardiac arrest patients receive standard advanced cardiac life support according to the 2015 AHA guideline, including chest compression, intubation, ventilation, defibrillation, drug administration, including epinephrine and antiarrhythmic drugs if indicated, in the emergency department.

A research associate generates a random sequence using Excel software, and assignment of participants to their respective groups will be undertaken by the principal investigator.

Arterial line insertion is performed within 6 minutes after randomization and diastolic blood pressure will be monitored.

If diastolic blood pressure is < 20 mmHg, drugs (vasopressin 40 IU or normal saline) will be administered for two times during CPR.

Arterial blood gas analysis will be analyzed for 5, 10, 15, and 20 minutes after arterial line insertion or termination of CPR.

End-tidal carbon dioxide concentrations is monitored in real time during CPR and recorded every minute.

The resuscitated patients receive standard post cardiac arrest care according to the 2015 AHA guideline.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic adult out-of-hospital cardiac arrest (OHCA) patients with non-shockable arrest rhythm

Exclusion Criteria:

* OHCA with terminal illness documented by medical record, under hospice care, with pregnancy, with pre-documented 'Do Not Resuscitate' card
* trauma patients
* age < 18 years old
* failed arterial line insertion within 6 minutes after randomization
* Extracorporeal cardiopulmonary resuscitation
* Time interval between arrest and ED arrival > 60 minutes
* ROSC within 6 minutes after ED arrival
* Diastolic Blood Pressure > 20 mmHg during resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Sustained return of spontaneous circulation (ROSC) | for 20 minutes after the time that participants had a palpable pulse
  CPCR result Achievement of sustained ROSC was declared when patients had a palpable pulse for more than 20 minutes.

SECONDARY OUTCOMES:
Improvement of arterial diastolic blood pressure assessed by arterial line | during CPR, every 10 seconds after arterial line insertion until the termination of CPR due to ROSC or death, whichever came first, assessed up to 30 minutes
  Successful adult resuscitation is more likely when diastolic blood pressure is > 25 to 30 mmHg.
  The 2015 AHA Guidelines for CPR and ECC recommend "trying to improve quality of CPR by optimizing chest compression parameters or giving vasopressors or both" if diastolic blood pressure is <20 mmHg.
  Investigators will record the hemodynamic monitor in real-time.
Improvement of end-tidal carbon dioxide concentrations assessed by capnography | during CPR, every one minute after endotracheal tube insertion until the termination of CPR due to ROSC or death, whichever came first, assessed up to 30 minutes
  End-tidal carbon dioxide concentrations during CPR are primarily dependent on pulmonary blood flow and therefore reflect cardiac output.
  Failure to maintain end-tidal carbon dioxide concentrations > 10 mmHg during adult CPR reflects poor cardiac output and strongly predicts unsuccessful resuscitation.
  Investigators will record the end-tidal carbon dioxide concentrations in real-time.
Improvement of acid-base status measured by blood-gas analysis | during CPR, 5, 10, 15, and 20 minute after arterial line insertion and termination of CPR
  Data are insufficient to make a conclusions, acid-base status can reflect the status of the ischemic insult on a cellular level. The changed of acid-base status during CPR may be associated with outcomes in cardiac arrest patients.
Improvement of lactate level measured by blood-gas analysis | during CPR, 5, 10, 15, and 20 minute after arterial line insertion and termination of CPR
  In previous studies, low lactate level was prognostic factors for favourable outcome after sustained ROSC.
  Lactate level can reflect the status of the ischemic insult on a cellular level.
Low level of neuron specific enolase level | 24, 48, and 72 hours after ROSC
  Low level of neuron specific enolase level is known as a prognostic indicator of neurologic outcome after cardiac arrest.
Good neurological outcome based on Cerebral Performance Categories Scale | checked at hospital discharge (participants will be followed for duration of hospital stay, an expected average of 4 weeks)
  CPC 1. Good cerebral performance: conscious, alert, able to work, might have mild neurologic or psychologic deficit. CPC 2. Moderate cerebral disability: conscious, sufficient cerebral function for independent activities of daily life. CPC 3. Severe cerebral disability: conscious, dependent on others for daily support because of impaired brain function. CPC 4. Coma or vegetative state: any degree of coma without the presence of all brain death criteria. CPC 5. Brain death: apnea, areflexia, EEG silence, etc.
  Good neurologic outcome is defined as CPC 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Won Young Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Chonnam National University Hospital, Gwangju
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh DK, Kim JS, Ryoo SM, Kim YJ, Kim SM, Hong SI, Chae B, Kim WY. Augmented-Medication CardioPulmonary Resuscitation (AMCPR) trial: a study protocol for a randomized controlled trial. Clin Exp Emerg Med. 2022 Dec;9(4):361-366. doi: 10.15441/ceem.22.367. Epub 2022 Nov 2. PMID 36318879